CLINICAL TRIAL: NCT04349722
Title: A Randomised Control Study: The Effect of Hyoscine-N-butylbromide (HBB, Buscopan) in Augmented Labour Among Primigravidae
Brief Title: The Effect of Hyoscine-N-butylbromide (HBB, Buscopan) in Augmented Labour Among Primigravidae
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Rahana Abd Rahman, Co-primary investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF-2019-521
Record Dates: First submitted 2020-04-12; First posted 2020-04-16 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Labor Long
Keywords: hyoscine; Duration of labour
MeSH Terms: interventions — Butylscopolammonium Bromide

STUDY DESIGN:
Intervention Model Description: Comparison between participants who receive hyoscine and those who do not.
Who Masked: Participant, Care Provider
Masking Description: Participants and care provider are blinded from the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyoscine (Active Comparator): Participants receive intravenous bolus of 1ml (20 mg) Hyoscine
  Interventions: Drug: Hyoscine Butylbromide
- Placebo (Placebo Comparator): Participants receive intravenous bolus of 1ml normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hyoscine Butylbromide — Intervention is given once a participant is in established labor
  Other Names: Buscopan
  Arms: Hyoscine
Other: Placebo — Intervention is given once a participant is in established labor
  Arms: Placebo

SUMMARY:
This study compares the duration of active phase of labour in women who received buscopan and those who don't.

DETAILED DESCRIPTION:
A randomised control study involving primigravida in labour who require pitocin augmentation. Once patient require augmentation, patient will be randomised into intervention group (receiving intravenous buscopan 1ml or 20mg) and control group (intravenous normal saline 1ml). Both fluids are colourless. The primary outcome is duration from augmentation to os fully. The secondary outcome are to look on mode of delivery particularly any caesarean section due to failure to poor progress, maternal side effect (dry mouth and tachycardia) and baby outcome (apgar score and neonatal intensive care unit admission)

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* Vertex presentation
* Term gestation (37-41w)
* Active phase of labor (4cm with regular contraction at least 2:10)
* Spontaneous labor
* Oxytocin augmentation
* Maternal height ≥150cm

Exclusion Criteria:

* Multiple pregnancies
* Previous uterine surgery
* Hypertensive disease in pregnancy
* Gestational diabetes on treatment
* Clinical estimation of fetal weight >3.8kg
* Induction of labor
* Meconium stained liquor
* Allergy to hyoscine
* Medical contraindication to hyoscine (i.e Myasthenia gravis, glaucoma, megacolon)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Labor length | Through study completion until delivery up to 12 hours
  Duration of labor

SECONDARY OUTCOMES:
Maternal age | At the time of recruitment
  Mean maternal age in years
Gestational age | At the time of recruitment
  Mean gestational age in weeks
Pre-pregnancy body mass index | At the time of recruitment
  Mean body mass index in kg/m2
First stage of labor | From onset of regular contraction to cervical dilatation of 10 cm up to 24 hours
  Mean duration of first stage of labor in hours
Second stage of labour | From cervical dilatation of 10cm until delivery of fetus
  Mean duration of second stage of labour in hours
Third stage of labour | From delivery of fetus until delivery of placenta
  Mean duration of third stage of labour in hours
Blood loss | Through study completion up to 42 days after delivery
  Mean blood loss in millilitres
Mode of delivery | Through study completion up to 12 hours
  Percentage of participants who delivered vaginally or via caesarean section
Analgesia | Through study completion until delivery up to 12 hours
  Percentage of women need analgesia
Pain score | Pre-intervention
  Mean pain score
Pain score 2 hours | From time of intervention up to 2 hours after
  Mean pain score at 2 hours
Pain score 4 hours | From time of intervention up to 4 hours after
  Mean pain score at 4 hours
Pain score 6 hours | From time of intervention up to 6 hours after
  Mean pain score at 6 hours
Neonatal outcome 1 minute | From delivery of neonate up to 1 minute after
  Mean apgar score at 1 minute
Neonatal outcome 5 minute | From delivery of neonate up to 5 minutes after
  Mean apgar score at 1 minute
Neonatal intensive care unit admission | From delivery of neonate up to 30 days
  Percentage of neonates require admission to neonatal intensive care unit admission
Side effects | Through study completion up to 42 days after delivery
  Percentage of participants who develop side effects to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aida Hani Mohd Kalok, Principal Investigator — National University Malaysia
Locations (1):
- National University Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia